CLINICAL TRIAL: NCT06836024
Title: Actazin (Kiwifruit Extract) Versus Polyethylene Glycol 3350 for Maintenance Therapy in Children With Constipation: a Feasibility Randomized Control Trial
Brief Title: A Trial of Actazin Versus PEG 3350 for Maintenance Therapy in Children With Constipation
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20240420-Kiwi
Record Dates: First submitted 2025-02-18; First posted 2025-02-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Constipation - Functional; Constipation; Constipation Aggravated
Keywords: Functional Constipation; Pediatric Constipation; Actazin; Kiwifruit Extract; Polyethylene Glycol 3350; Laxative Therapy; Randomized Controlled Trial; Feasibility Study; Non-Pharmacologic Treatment; Rome IV Criteria
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350; maltodextrin

STUDY DESIGN:
Intervention Model Description: Double dummy design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: each participant will receive both interventions, one will be active and the other will be placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Participants will receive Active Actazin chewable tablets and placebo maltodextrin powder resembling PEG 3350:
  1. Actazin oral chewable tablets with a starting dose of 600 mg (1 tablet) and can be titrated up to 2,400 mg (4 tablets).
  2. Placebo PEG 3350: Maltodextrin powder, administered in the same doses and manner as active PEG 3350 group.
  Interventions: Dietary Supplement: Actazin chewable tablet; Other: Maltodextrin (Placebo)
- Group 2 (Active Comparator): Participants will receive active comparator as PEG 3350 with a placebo chewable tablet resembling Actazin:
  1. PEG 3350 dissolved in 125-250 ml of cold water or juice (daily dose is age based: 4-5 years-2 tsp, 6-12 years-4 tsp; >13 years-5 tsp) and can be titrated by 1 tsp (3.7 grams) daily.57
  2. Placebo Actazin oral chewable tablets: Sorbitol-based placebo chewable tablets made by Pharma NZ Those tablets will have a similar appearance to active Actazin but will not taste the same. This is because the taste of Actazin is a non-altered natural kiwi taste. They will be administered in the same dose and manner as the active Actazin oral chewable tablets.
  Interventions: Drug: PEG 3350; Other: Chewable Tablet

INTERVENTIONS:
Dietary Supplement: Actazin chewable tablet — Actazin tablets are tableted non-GMO, freeze-dried, green kiwifruit powder from 100% New Zealand-grown green kiwifruit. Currently, kiwifruit extracts (such as Actazin), are marketed in Canada as a natural supplement. It is safe, bioavailable, and has been previously shown to be well tolerated at doses up to 2400 mg.
  Arms: Group 1
Drug: PEG 3350 — a commonly used over the counter laxative in north America. A stool softener.
  Arms: Group 2
Other: Chewable Tablet — Sorbitol-based placebo chewable tablets made by Pharma NZ. Those tablets will have a similar appearance to active Actazin but will not taste the same. This is because the taste of Actazin is a non-altered natural kiwi taste. They will be administered in the same dose and manner as the active Actazin oral chewable tablets.
  Arms: Group 2
Other: Maltodextrin (Placebo) — Maltodextrin powder, administered in the same doses and manner as active PEG 3350 group.
  Arms: Group 1

SUMMARY:
The goal of this pilot feasibility randomized controlled trial is to determine whether Actazin (kiwifruit extract) is a feasible and effective alternative to polyethylene glycol 3350 (PEG 3350) for maintenance therapy in children with functional constipation (FC). This study will include children aged 4 to 17 years who meet the Rome IV criteria for functional constipation.

The main questions it aims to answer are:

1. Is it feasible to conduct a definitive, multi-centre trial comparing Actazin to PEG 3350 in children with FC?
2. What are the within-group differences in clinical outcomes such as stool frequency, abdominal pain, and laxative use over a 4-week period?

Researchers will compare chewable Actazin tablets with placebo PEG 3350 powder to PEG 3350 powder with placebo Actazin tablets to see if Actazin is a viable non-pharmacologic natural health product alternative for treating FC.

Participants will:

Undergo an initial bowel cleanout using PEG 3350 and bisacodyl. Following, they will be randomized to one of two groups:

1. Actazin chewable tablets (titrate to effect: 600-2400 mg/day) + placebo PEG 3350
2. PEG 3350 (dose based on age and titratable to effect) + placebo Actazin chewable tablets Participants will take the assigned intervention daily for 4 weeks and complete a daily bowel diary recording stool frequency, consistency (Bristol Stool Scale), abdominal pain, and laxative use. They will have weekly follow-ups via phone or electronic survey to assess adherence, medication use, and adverse events.

Additionally, a bi-weekly follow-up will be conducted for an additional 8 weeks to track longer-term outcomes.

Outcomes:

Primary feasibility outcomes include consent rate, adherence to allocated intervention, and 4-week follow-up completion rate.

Secondary clinical outcomes include resolution of FC (Rome IV criteria), weekly stool frequency, abdominal pain episodes, use of rescue laxatives, and treatment palatability.

This study is being conducted at McMaster Children's Hospital and is funded by the Hamilton Academic Health Sciences Organization (HAHSO). Data collection will be managed using the Lumedi™ platform, and safety will be overseen by a Data Safety Monitoring Board (DSMB).

DETAILED DESCRIPTION:
This pilot feasibility randomized controlled trial aims to evaluate the feasibility and preliminary efficacy of Actazin (kiwifruit extract) versus polyethylene glycol 3350 (PEG 3350) as a maintenance therapy for children with functional constipation (FC). The study follows a double-dummy, quadruple-masked, single-centre design to ensure blinding of participants, caregivers, healthcare providers, and investigators.

The trial will enroll children aged 4 to 17 years diagnosed with functional constipation based on Rome IV criteria, recruited from the emergency department (ED) and outpatient clinics at McMaster Children's Hospital (MCH). The study will examine whether a larger, multi-centre trial is feasible based on recruitment rates, adherence to the intervention, and follow-up retention.

Study Design

This is a randomized, double-dummy, quadruple-masked feasibility trial evaluating Actazin against PEG 3350 for the maintenance management of pediatric FC. Sixty participants will be enrolled and randomized in a 1:1 ratio to either:

Intervention group:

Actazin chewable tablets (600 mg starting dose, titrated up to 2,400 mg daily) + placebo PEG 3350 powder Comparator group: PEG 3350 powder (age-based dose) + placebo Actazin chewable tablets Participants and caregivers, bedside clinicians, outcome assessors, and investigators will all be masked to the treatment allocation. The study will last 4 weeks, followed by an additional 8-week observational follow-up to assess longer-term adherence and clinical effects.

Randomization & Blinding:

Conducted using block randomization (blocks of 2, 4, or 6) through the Hamilton Health Sciences (HHS) Research Pharmacy. Participants will receive identically packaged drug kits containing either active treatment or placebo.

Data Collection & Monitoring Participants and caregivers will complete a daily bowel diary electronically. Weekly remote follow-ups (phone or electronic survey) will monitor adherence, medication use, and any adverse events.

The final statistical analysis will include descriptive and exploratory methods, reporting mean differences and confidence intervals for clinical outcomes.

Statistical Analysis Plan

Feasibility analysis will be based on progression criteria:

If all feasibility outcomes meet the predefined thresholds, the trial will proceed to a definitive multi-centre RCT. If one or more outcomes fall below feasibility thresholds, protocol modifications will be considered. Clinical outcomes will be analyzed using linear regression (continuous variables) and logistic regression (binary outcomes). Adverse event rates will be compared between groups using Fisher's exact test. No formal hypothesis testing for efficacy will be conducted, as this is a pilot feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 to 17 years, inclusive; minimum age of 4 years to ensure toileting skills have been acquired and ability to chew and swallow tablets safely.
2. Fulfill Rome IV diagnostic criteria for FC;60 Must include ≥2 of the following occurring at least once per week for a minimum of 1 month: (i) ≤2 SBMs/ week; (ii) ≥1 episode of fecal incontinence/week; (iii) retentive posturing; (iv) painful or hard bowel movements; (v) presence of a large fecal mass in the rectum (rectal, abdominal or radiographic exam) and (vi) history of large-diameter stools that can obstruct the toilet.
3. Participant and their caregivers agree to exclusively use the laxatives provided as part of the trial for a 4-week period, and refrain from using any additional PEG 3350 or kiwifruit/kiwifruit extracts outside of the trial products.

Exclusion Criteria:

1. Organic causes of constipation (e.g., celiac disease, Hirschsprung's disease, spina bifida, anorectal malformations)
2. Prior enrollment in trial
3. Not toilet trained; significantly different FC phenotype than toilet trained children
4. Any known hypersensitivity to kiwifruit, latex, Actazin or PEG 3350
5. Chronic health conditions (e.g., urolithiasis, ureteropelvic junction obstruction, sickle cell, cerebral palsy, hepatic, hematopoietic, renal, endocrine, or metabolic diseases) that could potentially confound the results of the study
6. Prior abdominal surgery involving the luminal GI tract, except hernia repairs
7. Concomitant use of drugs that are known to affect GI motility (e.g., opioids, domperidone, linaclotide)
8. Prior neuropsychiatric or pervasive developmental disorders such as severe non-verbal ASD, major psychiatric disorders (bipolar disorder, schizophrenia, major depression)
9. Refractory or severe FC that failed to respond to PEG 3350 and/or require combination of several laxative therapies, manual disimpaction, use of any nerve stimulation or antegrade enemas through a cecostomy or an appendicostomy
10. Absence of a parent/guardian for children who are not mature minors
11. Inability to obtain consent due to a language barrier and the absence of language translator in person or by a phone translation service available in the ED

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Consent Rate | 18 months
  Total number consented / Total number eligible and approached for consent
4-week Follow up rates | 18 months
  Total number of participants who did not complete the 4-week outcome
Adherence to allocated intervention | 18 months
  Total number of participants who received the intervention they were allocated and did not cross over / Total number of participants

SECONDARY OUTCOMES:
Recruitment rate | 18 months
  Number of participants recruited/month
Eligibility criteria | 18 months
  Proportion who are being assessed and treated for constipation, but do not meet Rome IV criteria
Completion of daily bowel diary | 18 months
  Number of missing items on the data collection form / total number of variables collected
Compliance rate | 18 months
  Number of days participants took laxative / 28 days
Palatability | 18 months
  Visual analogue scale with 10 facial hedonic features (0-10)

OTHER OUTCOMES:
ROME IV criteria | 18 months
  FC resolution (not meeting Rome IV FC criteria) at 28 days (+/-3 days) of treatment
proportion with clinical resolution of functional constipation | 18 months
  weeks 1-3, not meeting Rome IV FC criteria
weekly frequencies of the itemized items in Rome IV criteria | 18 months
  Spontaneous Bowel Movements (SBMs) - Frequency per week Episodes of Fecal Incontinence - Number of occurrences per week Retentive Posturing (Withholding Behaviors) - Number of episodes per week Painful or Hard Bowel Movements - Number of painful stools per week Presence of a Large Fecal Mass in the Rectum - Identified through clinical exam (weekly assessment) History of Large-Diameter Stools that Can Obstruct the Toilet - Caregiver-reported frequency per week
Stool consistency | 18 months
  Daily Bristol Stool Scale score (1 to 7) Type 1: Separate hard lumps (like nuts, hard to pass) Type 2: Sausage-shaped but lumpy Type 3: Sausage-shaped with cracks on the surface Type 4: Smooth, soft, and sausage-like Type 5: Soft blobs with clear-cut edges (easy to pass) Type 6: Mushy, fluffy pieces with ragged edges Type 7: Completely liquid, no solid pieces
Abdominal pain | 18 months
  daily frequency of abdominal pain episodes; pain frequency will be determined by the number of pain episodes with ratings of ≥1/10 on the verbal numerical rating scale over a 4-week diary (0 is no pain, 10 is the worst pain ever)
Rescue laxatives | 18 months
  frequency of weekly use of rescue laxatives
Bloating | 18 months
  child report of daily presence or absence of bloating (defined as a sensation of fullness of the abdomen with or without gurgling or rumbling noises, excessive flatulence or visible swelling of the abdomen)
School or camp or daycare abscence | 18 months
  number of days absent from school/daycare/summer camp due to constipation

CONTACTS AND LOCATIONS:
Overall Officials: Elyanne Ratcliffe, MD, Principal Investigator — Hamilton Health Sciences Corporation; Mohamed M Eltorki, MBChB, MSc, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request.